CLINICAL TRIAL: NCT06763783
Title: Vaccination in Patients With Inflammatory Rheumatic Diseases. The Impact of Anti-rheumatic Treatments on the Immunogenicity of Herpes-zoster Vaccine (Shingrix) and Protection Against Infection (HZ-REUMA)
Brief Title: Vaccination Against Herpes Zoster in Patients With Inflammatory Rheumatic Diseases
Acronym: HZ-REUMA
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2023-506230-71-01
Record Dates: First submitted 2024-12-18; First posted 2025-01-08 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-12

CONDITIONS: Systemic Vasculitis; Spondylarthropathies; Psoriatic Arthritis; Scleroderma; Polymyalgia Rheumatica (PMR); Juvenile Chronic Arthritis; Polyarthritis; SLE; Giant Cell Arteritis (GCA)
Keywords: herpes zoster; vaccine response; inflammatory rheumatic disease
MeSH Terms: conditions — Systemic Vasculitis; Spondylarthropathies; Arthritis, Psoriatic; Scleroderma, Diffuse; Polymyalgia Rheumatica; Arthritis, Juvenile; Arthritis; Giant Cell Arteritis; Herpes Zoster | interventions — Vaccination

STUDY DESIGN:
Intervention Model Description: patients with different rheumatic diseases receiving different immunosuppressive treatments (active group) and patients with different rheumatic diseases without immunosuppressive treatment (control) receive 2 doses of subunit vaccine against herpes zoster (Shingrix). Vaccine response between the two groups will be compared
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- all participants will be vaccinated with two doses Shingrix vaccine (Other): all participants will be vaccinated but the difference in the antibody and T cells responses to vaccination will be compared between the grupp of patients treated with immunomodulating drigs and patients not receiving such treatments
  Interventions: Drug: Shingrix; Drug: vaccination with 2 doses of Shingrix vaccine

INTERVENTIONS:
Drug: Shingrix — all participants vaccinates with two doses of Shingrix vaccine
Drug: vaccination with 2 doses of Shingrix vaccine — all participants will receive vaccination with 2 doses of Shingrix vaccine. The response to caccine will be compared bitween patients treated with immunosupressive drugs and these not receiving immunosuppresive treatment

SUMMARY:
The purpose of HZ-REUMA study is explore vaccine response and protection against shingles (herpes zoster, HZ) after vaccination with two doses of Shingrix in immunosuppressed patients with inflammatory rheumatic diseases (IRD) compared to immunocompetent patients with IRD (controls).

Hypothesis:

The immunological disturbance as part of the rheumatic disease in combination with different immunomodulating treatments may impair vaccine response to non-live HZ vaccine (Shingrix) and thereby lead to an insufficient protection against infection.

Primary objective (outcome)

1. The impact of modern anti-rheumatic treatments including synthetic disease modifying anti-rheumatic drugs (DMARDs) such as methotrexate and different biological treatments (anti-TNF, anti IL6r, anti-IL12/23/17, anti-CD20, anti-BlyS, anti-INFERON treatment, or targeted DMARDs (JAK-inhibitors) on antibody response elicited by two doses of subunit vaccine against herpes zoster (HZ) administrated 1-2 months apart in patients with IRD.

   Secondary outcomes
2. The numbers and frequency of antigen specific CD4 2+ T cells expressing ≥2 or more activation markers (TNFalpha, INF-gama, interleukin-2 or CD40ligand)
3. Long-term immunogenicity of two doses of Shingrix in immunosuppressed patients with IRD measured 3 and 5 after vaccination
4. the tolerability of the vaccine, the impact on existing rheumatic disease, and possible association with onset of new autoimmune diseases
5. if vaccination against herpes zoster protects against infections in patients with inflammatory rheumatic diseases

Study Population Adult patients (18 years and older) with a clinically diagnosed inflammatory rheumatic disease and regularly followed at Skåne University Hospital, section for rheumatology in Lund/Malmö, Sweden are eligible for the study and will be offered vaccination free of charge. Control group comprises adult individuals with known inflammatory rheumatic disease without immunosuppressive treatment except for low dose prednisone (max 5 mg daily) .

Inclusion criteria:

* age ≥18 years (patients)
* regular follow up at Skåne University Hospital, section for rheumatology Lund/Malmö due to an inflammatory rheumatic disease (patients)
* receive active treatment with disease modifying anti-rheumatic drugs (DMARDs) such conventional synthetic (cs), biologic (b) or targeted synthetic (ts) DMARDs or patients without active immunosuppressive treatment (controls)

Exclusions criteria

* age <18 years (patients)
* pregnancy (women of childbearing potential, WOCBP, are not excluded since all patients using DMARDs are advised to use a safe and effective contraceptive method)
* allergy/intolerability of any component in the vaccine
* active infection inclusive herpes zoster (shingles)
* received Shingrix vaccine previously
* ongoing treatment with any immunosuppressive drug for the other diseases Target enrolment/sample size: 240. Study start date: December, 17 2024- June 30, 2029

DETAILED DESCRIPTION:
Patients with inflammatory rheumatic diseases (IRD) such as rheumatoid arthritis (RA), SLE, spondyloarthropathies, systemic vasculitis or systemic sclerosis (Granulomatosis with polyangiitis, GPA; Eosinophilic granulomatosis with polyangiitis, EGPA, Giant Cell Arteritis, GCA), systemic sclerosis or other inflammatory systemic disease) have an increased morbidity and mortality in infections. These infections include the numerous vaccine-preventable diseases such as herpes zoster (HZ). Vaccination is a cost-effective measure to prevent an infection. However, several studies have reported an impaired response to common vaccinations among immunosuppressive patients with IRD. The underlying mechanisms are not entirely known. The Centre for Disease Control (CDC) Advisory Committee for Immunization Practice (ACIP) as well as the European League Against Rheumatism (EULAR) and Swedish authorities (The Public Health Agency of Sweden) recommend vaccination against HZ to the risk groups. Majority of patients with IRD are treated with potent immunosuppressive drugs and thereby belong to the target group for HZ vaccine. Data on the immunogenicity, tolerability of a non-live, subunit vaccine against HZ (Shingrix) among immunosuppressed patients with IRD is limited. The overall aim of this research project is to study antibody and T cells response and tolerability of two doses of subunit HZ vaccine (Shingrix) in immunosuppressed patients with IRD compared to IRD patients without active immunosuppressive treatment (with exception for prednisolone orally in a maximal daily dose of 5 mg).

Hypothesis The immunological disturbance as part of the rheumatic disease in combination with different immunomodulating treatments may impair antibody and T cells vaccine response but vaccination is still expected to generate a "satisfactory immune response".

Main objective (outcome)

To study:

1. The impact of modern anti-inflammatory treatments including synthetic disease modifying anti-rheumatic drugs (DMARDs) such as methotrexate and different biological treatments (anti-TNF, anti IL6r, anti IL12/23/17, anti CD20, JAK-inhibitors, anti-BlyS, anti-INF, or targeted DMARDs (JAK-inhibitors) on antibody response elicited by two doses of subunit vaccine against herpes zoster (HZ) administrated 1-2 months apart in patients with IRD Secondary objectives (outcomes)
2. The numbers and frequency of antigen specific CD4 2+ T cells expressing ≥2 or more activation markers
3. Long-term immunogenicity (measured as GML of anti-gE antibodies and numbers and frequency of antigen specific CD4 2+ T cells expressing ≥2 or more activation markers 3 and 5 years after vaccination with two doses of Shingrix vaccine
4. the tolerability of the vaccine including the impact on existing rheumatic disease (increased activity/flare/possible association with onset of new potential immune-mediated diseases (pIMD) or herpes zoster case during the study period, see the enclosed algorithm.
5. if vaccination against herpes zoster protects against infections in patients with inflammatory rheumatic diseases

Safety assessments and safety reporting -At vaccination (visit 1 and 2) when the first and second vaccine doses are administrated each participant will receive oral information on the common adverse events (AE), adverse drug reactions (ADR) and serious adverse events (SAE). AEs/ADRs will be assessed and reported using the GSK global safety document.

Safety Reporting Institution/Investigator is solely responsible for reporting all Adverse Events and Serious Adverse Events to regulatory authorities, investigators, IRBs or IECs, and GSK, as applicable, in accordance with national regulations in Sweden where the study is conducting.

Severity of Event

1. (mild)= An AE which is easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities.
2. (moderate) = An AE which is sufficiently discomforting to interfere with normal everyday activities.
3. (severe)= An AE which prevents normal, everyday activities. Such an AE would, for example, prevent attendance at work/school and would cause the participant to seek medical advice.

Collection and Reporting of AEs & SAEs Study patients will be instructed to contact the study staff if any serious or unexpected adverse event occurs. Reported AE's will be recorded in detail in an AE case report form. Adverse events will be identified with patients during study visits. Any adverse events will be discussed with the PI and will be reviewed to determine whether a change in protocol is necessary.

All adverse events and serious adverse events should be recorded on the Adverse Event Log, Serious Adverse Event Log, and in Data Management system, within 24 hours.

Fatal and Life Threatening SAEs within 24 hours of the investigator's observation or awareness of the event.

All other serious (non-fatal/non-life threatening) events within 4 calendar days of the investigator's observation or awareness of the event.

All pregnancy events within 4 calendar days of the investigator's awareness of the event. All pIMDS or exacerbation of pIMDS events within 7 calendar days of the investigator's observation or awareness of the event.

In addition, each participant is provided with a written questionnaire on the possible effects from the vaccination (AE, ADR or SAE) with instructions how to record them and a telephone number to the research nurse in case of more serious side effects or emergency department (life-threatening effects). In case of reactivation of HZ infection all participants are encouraged to contact the research nurse for an extra visit för VZV PCR or serological response and anti-viral treatment according to algorithm.

PI will report AEs/SAEs to the authorities, IRBs/IECs as appropriate. AEs will be graded as mild, moderate, severe and life threatening. All SAEs, pIMDs will be reported to GSK within 24 hours to the GSK Safety mailbox: ogm28723@gsk.com.

All ADRs that are both serious and unexpected are subject to expedited reporting by the PI. All serious effects will be reported to the authorities as required i.e. effects no later than 15 calendar days after first knowledge (serious) and as soon as possible but no later than 7 calendar days after first knowledge (lethal/life-threatening adverse/unexpected effects. The GSK AE case report form will be used for reporting ARDs and SAEs.

Additional safety endpoints: an exacerbation of pre-existing rheumatic disease accessed by the rheumatologist/ PI/sub-investigators, or an onset of other auto-immune conditions (see list) requires assessment by the PI and will be reported, recorded in details and followed until resolved.

Inclusion criteria:

* age ≥18 years
* has diagnosed an inflammatory rheumatic disease
* has a regular follow up at Dept of rheumatology, Skåne University Hospital Lund/Malmö
* receives active treatment with disease modifying antirheumatic drugs (DMARDs) such conventional synthetic (cs), biologic (b) or targeted synthetic (t) DMARDs [patients in the study] or no active treatment with s/b/t DMARDs with exception of daily prednisolone dose of max 5 mg [controls in the study]
* a safe preventive method for women before menopause
* is able to sign a consent

Exclusion criteria:

* age <18 years
* pregnancy (women of childbearing potential, WOCBP need to declare the using a safe contraceptive method)
* allergy/intolerability of any component in the vaccine
* acute disease and/or fever at the time of vaccination. Fever is defined as temperature ≥ 37.5°C by oral route. (The preferred route for recording temperature in this study will be oral). Subjects with a minor illness (such as mild diarrhea, mild upper respiratory infection) without fever may be enrolled at the discretion of the investigator
* received Shingrix vaccine previously
* ongoing treatment with any immunosuppressive drug for other disease with exception for prednisolone in a daily dose corresponding max 5 mg before the inclusion
* participates or has participated in the other interventional clinical study within 3 months before the inclusion
* taking concurrently medication which is not approved in EU

Study Design and Methods

* Patients with inflammatory rheumatic disease receiving active anti-rheumatic treatment (see inclusion criteria) are offered to participate at routine visit at the out- patient clinic
* Controls -patients with known rheumatic disease not taking any immunosuppressive drugs for any disease with exception for prednisolone in a daily dose corresponding max 5 mg
* All participant receives a unique, individual study code (HZ-REUMA001, HZ-REUMA002, HZ-REUMA003, ….) The study code and all study documentation are stored at a safe place at the department and only PI and sub-investigator (HK) have access to them. In case of safety issues during the study, PI and sub-investigator may upon request provide all data collected on the actual case, to healthcare providers .

At vaccination (visit 1) the physical examination is performed by a rheumatologist and data on disease and treatment characteristics, anti-rheumatic treatments and other concomitant treatments including previous vaccinations and history of varicella or HZ (study questionnaire), co-morbidity (Charlson Comorbidity Index (CCI), smoking habits (questionnaire), physical function (health assessment questionnaire, HAQ;), EQ5D are collected.

-Patients reported outcome (HAQ, EQMD) are registered in the Swedish rheumatology registry (SRQ) which is a part of a routine care.

Blood Sampling

Blood will be collected pre-vaccination, 4-6 weeks post-dose 2, thereafter 3 years, and 5 years (see schedule of activities).

* Blood samples (6 ml blood) are collected for the analyses of inflammatory markers (CRP, ESR, Hb, total leucocyte count, and differential leucocyte count, ALT and creatinine) performed immediately at the local biochemical lab (1 ml). Remaining 5 ml are stored as a serum samples at -80C in the biobank at the rheumatology department and will be used for future analyze of serological response (IgG antibodies against glycoprotein E). This analysis (ELISA) will be performed simultaneously on all pre - and postvaccination samples at three different occasions i.e. 4-6 weeks following the second vaccine dose, after 3 and 5 years follow ups, respectively. This analysis will be performed in collaboration with Professor Tomas Bergström at Institution for virology, Sahlgrenska academy, Gothenburg (Sweden). GSK will share some information about the anti-gE ELISA developed by GSK.
* Additional 30 ml of peripheral blood will be collected maximally few hours before shipping to Institution for virology, Sahlgrenska academy, Gothenburg (Sweden) where the analyses of vaccine specific T cells response will be performed. Blood samples are collected into a tube containing the standard anticoagulant (sodium heparin) and labelled with the identifier (study code, date and time), gently rocked approximately every 2 hours and maintained in room temperature (17-24 ◦C) during the transportation. The samples are processed and analyze as soon as possible after the arriving to the lab using the standardized protocol. The analysis includes the measuring of number and function of antigen specific of CD4 + positive T-cells expressing at least 2 activity markers (for example TNFalpha, INF-gamma, interleukin-2 or CD40ligand) using flowcytometry

Statistical Plan and data analysis The study population comprise at least 240 individuals who have received two vaccine doses, whose blood samples have been collected before vaccination and the second vaccine dose. Of these, 190 are patients and 50 controls (patients not receiving any immunosuppressive treatment). In order to ensure the number of participants who fulfil these criteria approximately 10% additional participants (both patients and controls) will be recruited.

Patient groups will be further stratified in two groups, according to either immunosuppressive treatment or diagnosis . Geometric mean antibody levels, GML after vaccination compared to pre-vaccination GML. The percentage of responders (defined as ≥ 4-fold increase in pre-vaccination antibody levels) are assumed to be 99,99% and 80% in control respectively. In order to compare % responders in controls (n=50) and patient group (n=190) with a planned sample size we will have an 80% power to detect 20% unit difference with 5% significance and two sided hypothesis.

Power calculation Two-sided confidence interval (%) 95 Number of exposed immunosuppressed patients 190 Risk of disease among exposed (%) 80 Number of non-exposed 50 Risk of disease among non-exposed (%) 99 Risk ratio detected 0.81

Power based on:

Normal approximation 90.78% Normal approximation with continuity correction 86.38% Percentage of participants seropositivity and seroconversion (after two vaccine doses) will be calculated and compared between two groups. GML before and after will be compared between the groups.

In addition, statistical comparation will be performed with patients receiving only one vaccine dose using appropriate statistical analysis (depending on the number of such cases).

Details around stratification of patients:

* Further stratification of patients will be done into following groups csDMARDs (such as methotrexate, azathioprine, sulfasalazine), bDMARDs (such as anti-TNF, anti-IL6r, anti-CD20, abatacept) and tsDMARD (JAK-inhibitors). Vaccine response in each of these 3 groups can be compared to controls
* Logistic regression analysis adjusted for baseline disease and treatment characteristics including usage of oral prednisolone will be performed to study the impact of on the vaccine response.

Significance Results from this project will be used to support recommendations on vaccination against HZ in immunosuppressed patients known to be at an increased risk of HZ and its complications.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (age 18 years and older) with clinically diagnosed inflammatory rheumatic disease who are regularly followed at Skåne University Hospital, section for rheumatology in Lund and Malmö, Sweden are eligible for the study and will be offered vaccination with 2 doses of Shingrix free of charge. Control group comprises adult patients with inflammatory rheumatic diseases not receiving immunosuppressed drugs but receive 2 doses of Shingrix.

* age ≥18 years
* has diagnosed an inflammatory rheumatic disease
* has a regular follow up at Dept of rheumatology, Skåne University Hospital Lund/Malmö
* receives active treatment with disease modifying antirheumatic drugs (DMARDs) such conventional synthetic (cs), biologic (b) or targeted synthetic (t) DMARDs [patients in the study] or no active treatment with s/b/t DMARDs with exception of daily prednisolone dose of max 5 mg [controls in the study]
* a safe preventive method for women before menopause
* is able to sign a consent

Exclusion Criteria:

* age <18years
* pregnancy (women of childbearing potential, WOCBP need to declare the using a safe contraceptive method)
* allergy/intolerability of any component in the vaccine
* acute disease and/or fever at the time of vaccination. Fever is defined as temperature ≥ 37.5°C by oral route. (The preferred route for recording temperature in this study will be oral). Subjects with a minor illness (such as mild diarrhea, mild upper respiratory infection) without fever may be enrolled at the discretion of the investigator
* received Shingrix vaccine previously
* ongoing treatment with any immunosuppressive drug for other disease with exception for prednisolone in a daily dose corresponding max 5 mg before the inclusion
* participates or has participated in the other interventional clinical study within 3 months before the inclusion
* taking concurrently medication which is not approved in EU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2034-06-30 (Estimated)

PRIMARY OUTCOMES:
Pre-and post-vaccination anti-gE antibody levels (geometric mean antibody levels, GML) in patients and controls | before vaccination and 4-6 vecks after the second vaccine dose
  Measurement of pre-and post-vaccination anti-gE antibody (g/L) in patients and controls which will be used for calculating the proportion of individuals in different treatments group and controls with ≥4-fold increase in anti-gE antibody measured 4-6 weeks following the second vaccine dose (vaccine response rate)

SECONDARY OUTCOMES:
Number and function of antigen (vaccine) specific T cells | before vaccination and 4-6 weeks after second vaccine dose
  Number and function of vaccine specific T cells before vaccination and 4-6 weeks after second vaccine dose which express ≥2 or more activation markers in all participants
long-term immunogenicity | 3 and 5 years after inclusion
  Measurement of postvaccination antibody levels (g/L) after 3 and again after 5 years from inclusion in all participants which will be used to calculate the proportion of individuals with ≥4-fold increase in antibody levels compared to pre-vaccination antibody levels in patients and controls, respectivelly.
the tolerability of the vaccine | from inclusion to 6 months after the inclusion of last patient
  number of patients and controls with moderate, serious and life threatening adverse effects as well as number of herpes zoster infections after the first, and after the second vaccine dose
number of HZ infections in vaccinated individuals | from 1 months after the second vaccine dose to the study end 2034
  number of herpes zoster infections in vaccinated patients

CONTACTS AND LOCATIONS:
Locations (1):
- Skåne University Hospital, section for rheumatology, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: after the study completition